CLINICAL TRIAL: NCT03637777
Title: Characterization of the Reproductive Tract and Gastrointestinal Tract Microbiome and Its Association With Pregnancy Outcomes Following Frozen Embryo Transfer
Brief Title: The Human Microbiome and IVF Outcomes
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2017-03
Record Dates: First submitted 2018-08-09; First posted 2018-08-20 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, urine, buccal, cervical, vaginal, rectal, semen, embryo transfer catheter tip
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 16S rRNA gene sequencing — Specimens collected from patients will be used for next generation sequencing of the bacteria-specific 16S rRNA gene

SUMMARY:
Patients and partners undergoing an autologous IVF cycle will be recruited to participate in this prospective observational study investigating the microbiome and its association with IVF pregnancy outcomes. During the the controlled ovarian hyperstimulation cycle as well as the frozen embryo transfer cycle, a number of specimens will be collected for next generation sequencing of 16S rRNA to evaluate the microbiome profile of the reproductive and gastrointestinal tracts. Data on pregnancy outcomes will be collected prospectively and evaluated to identify associations with the microbiome.

DETAILED DESCRIPTION:
PURPOSE OF STUDY

To characterize the microbiome of the female reproductive tract and gastrointestinal tract as well as the male reproductive tract in patients and partners undergoing IVF and determine if there are any associations with pregnancy outcomes.

The Clinical Problem

The microbiome of the reproductive tract and its association with reproductive outcomes is a topic of evolving interest. Alterations in the vaginal microbiome have been linked to obstetric complications including miscarriage and preterm birth. More recent data have emerged linking the vaginal microbiome to assisted reproductive technology (ART) outcomes. A prospective observational study consisting of 30 patients who had swabs collected at various time points during the in vitro fertilization-embryo transfer (IVF-ET) cycle for sequencing of the 16S ribosomal RNA gene concluded that the species diversity of the vaginal microbiome distinguished women who had a live birth from those who did not with increased diversity being associated with poorer outcomes; however, the patient population was heterogeneous and small.

Limited information is available regarding the microbiome of the upper genital tract and its association with reproductive outcomes, particularly in the setting of ART. Studies done solely for the purpose of characterizing the upper genital tract microbiome have relied on hysterectomy specimens to assess colonization, thus precluding evaluation of any association with reproductive outcomes. Perhaps the first study to investigate the association between the microbiome of the upper reproductive tract and ART outcomes utilized culture-based technology on embryo transfer catheter tips. However, this study utilized culture-based technology, with only four major bacteria were reported. Subsequent studies have highlighted the limitations of culture-based technology, namely that it is reliant upon successful culture, often resulting in an underestimate of the diversity of organisms.

As sequencing-based technology has gained popularity and limitations of culture-based technology have become more evident, there has been an increased interest in using sequencing to characterize the microbiome. One recent study utilized next-generation sequencing (NGS) based technology on embryo transfer catheter tips to evaluate the bacteria specific 16S ribosomal gene for characterization of the upper genital tract microbiome in patients undergoing embryo transfer. Although it served as proof of concept for this method of characterizing the microbiome, the limited sample size did not permit any conclusions to be drawn regarding its association with reproductive outcomes. A subsequent study utilizing sequence-based technology examined endometrial fluid and vaginal aspirate samples in 35 women in the cycle prior to IVF and found that the presence of non-Lactobacillus-dominated microbiota in the endometrium was associated with significant decreases in implantation, ongoing pregnancy and live birth.

Although there is some data linking reproductive health and the microbiome of the female reproductive tract, less information exists regarding its association with the microbiome of the male reproductive tract. One cross-sectional study examining the microbial colonization of semen demonstrated an association with semen parameters. Another study which examined vaginal and seminal cultures on 951 couples undergoing IVF found that positive bacterial cultures from both the vagina and semen decreased clinical pregnancy rate and increased miscarriage rate more than vaginal infection alone. The microbiome of the male reproductive tract warrants further investigation in this setting.

The gastrointestinal tract microbiome plays a major role in human health and disease, with many documented associations to disease states such as obesity, diabetes, and gastrointestinal disorders. Recent data suggests that alterations in gastrointestinal tract microbiota are associated with preterm labor. The urinary tract microbiome has been similarly studied and linked to multiple disease states such as urinary incontinence and chronic prostatitis.

To date, there are no published studies that examine the association of the gastrointestinal tract microbiome or urinary microbiota with pregnancy outcomes following IVF.

The human microbiome is thought to modulate the immune system and the presence of systemic inflammation. There is a growing interest in the association of chronic systemic inflammation and reproductive disorders. A number of biomarkers that reflect chronic systemic inflammation have been identified. Interleukin-6 (IL-6) is one such biomarker that has documented associations with PCOS, endometriosis, and infertility. Such biomarkers have not yet been studied in association with pregnancy outcomes following IVF.

The objective of this research is to perform a large-scale prospective observational study seeking to characterize the microbiome of the female reproductive tract (both upper and lower) at different time points in patients undergoing IVF. Furthermore, we plan to examine the female gastrointestinal tract microbiome, female urinary microbiota, and the microbiome of the male reproductive tract by collecting targeted specimens during patients' treatment cycles. Lastly, we will evaluate female and male serum for biomarkers of inflammation. We aim to identify any associations with pregnancy outcomes that may serve as a basis for a subsequent interventional study.

RESEARCH PROPOSAL

A. Location of Study:

Reproductive Medicine Associates of New Jersey

B. Study Population:

All patients initiating an autologous IVF cycle at our center will be reviewed for inclusion. Up to 1000 patients will be enrolled.

Major Inclusion Criteria: The following are major inclusion criteria:

1. Patients initiating an autologous IVF cycle
2. Patient age 18-45; partner age 18-60
3. Partner planning to provide fresh semen sample on day of oocyte retrieval
4. Patients planning to undergo preimplantation genetic screening (PGS) of embryos with single embryo transfer (SET)

Major Exclusion Criteria: The following are exclusion criteria:

1. > 1 prior failed IVF cycle
2. Third party reproduction
3. Planning to bank embryos
4. Partner using cryo sperm or surgical sperm on day of retrieval
5. Male or female partner antibiotic use within 1 month of IVF cycle start
6. Mullerian anomalies, excluding arcuate uterus
7. Submucosal fibroids
8. History of uterine surgery, excluding polypectomy, D&C, and Cesarean section
9. Communicating hydrosalpinx without plans for surgical correction prior to embryo transfer

C. Study Procedures:

Experimental Design

The proposed study is a prospective observational study which seeks to characterize the microbiome of the female reproductive tract at various time points during an IVF cycle and determine if there are any differences in the microbiome with respect to pregnancy outcomes. In addition, samples will be collected to evaluate the microbiome of the female gastrointestinal tract, female urinary microbiota, the male reproductive tract and biomarkers of systemic inflammation.

Study Related Clinical Procedures and Analyses

All patients initiating an autologous IVF cycle at our center will be reviewed for inclusion. Patients who meet study criteria will be contacted for possible enrollment. Once enrolled, patients and partners will be consented to participate in the study. They will proceed with treatment according to routine protocol and specimens will be collected for evaluation of the microbiome at designated time points.

The only study-related procedures that deviate from routine care will be the collection of specimens to be used for characterization of the microbiome and systemic inflammation at several time points throughout their care:

* Female

  * During the fresh IVF cycle: An additional tube of blood will be collected from the female partner at the time of a routine blood draw for cycle monitoring.
  * Day of oocyte retrieval: A mid-stream urine sample will be provided by the female partner on the morning of oocyte retrieval. Cervical, vaginal, buccal and rectal swabs will be collected from the patient while under sedation just prior to the oocyte retrieval procedure.
  * During the FET cycle: An additional tube of blood will be collected from the female partner at the time of a routine blood draw for cycle monitoring.
  * Mid-proliferative scan during the first FET cycle: After a minimum of 8 days of estrogen exposure, a second set of cervical and vaginal swabs will be collected immediately prior to the patient's scheduled ultrasound.
  * Day of FET: When the patient presents for embryo transfer, a third set of cervical and vaginal swabs will be collected immediately prior to performing the embryo transfer. In addition, the most distal 5 mm portion of the transfer catheter will be collected after the embryo has been transferred.
* Male

  * During the fresh IVF cycle: One tube of blood will be drawn from the male partner.
  * Day of oocyte retrieval: A swab will be collected from the fresh semen specimen provided by the partner prior to any processing.

Blood will be allowed to clot prior to centrifugation. The specimens will be aliquoted and transferred to a -80°C for storage. They will subsequently be thawed as needed to analyze biomarkers of systemic inflammation. Remaining aliquots will be stored for potential future studies.

All other specimens will undergo cell lysis, DNA purification, and next-generation sequencing of the bacteria specific 16S ribosome gene according to previously published protocols.

Cycle outcomes will be recorded according to routine practice.

D. Risk/Safety Information:

The main risks of the blood draws are discomfort, bleeding, and bruising. All attempts will be made to coordinate collection of study blood with routine blood draws performed as part of the patient's clinical care. The main risk of vaginal/cervical swab collection is discomfort. Collection of the buccal and rectal swabs will be done under anesthesia at the time of the oocyte retrieval and therefore does not carry this risk. Collection of the mid-stream urine sample will be done when the patient empties her bladder prior to oocyte retrieval and does not pose any additional risks. Collection of the semen specimen does not involve any additional risk as the partner is providing a specimen as part of the treatment plan and the swab is collected after provision of the specimen. Collection of the transfer catheter tip does not involve any additional risk as it is performed after the embryo transfer is complete and does not directly involve the patient.

E. Data Management:

Statistical evaluation of the results

The microbiome at the various time points will be compared for patients with an ongoing pregnancy (as defined by presence of a fetal heartbeat at time of discharge) and those without. To characterize the diversity of samples, two alpha diversity metrics will be utilized: the Shannon diversity index (SDI) and chao1.

Study Length Timeline - 25 months

1. Time to recruit the study population - 12 months
2. Timeline for each individual participating in the study, from enrollment to delivery (if pregnant) - 10 months
3. Statistical analysis and manuscript preparation - 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients initiating an autologous IVF cycle
2. Patient age 18-45; partner age 18-60
3. Partner planning to provide fresh semen sample on day of oocyte retrieval
4. Patients planning to undergo preimplantation genetic screening (PGS) of embryos with single embryo transfer (SET)

Exclusion Criteria:

1. > 1 prior failed IVF cycle
2. Third party reproduction
3. Planning to bank embryos
4. Partner using cryo sperm or surgical sperm on day of retrieval
5. Male or female partner antibiotic use within 1 month of IVF cycle start
6. Mullerian anomalies, excluding arcuate uterus
7. Submucosal fibroids
8. History of uterine surgery, excluding polypectomy, D&C, and Cesarean section
9. Communicating hydrosalpinx without plans for surgical correction prior to embryo transfer

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients and partners undergoing IVF
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Live birth | 10 months
  Delivery of a live infant

SECONDARY OUTCOMES:
Ongoing pregnancy | 2 months
  Presence of fetal heart beat at 8 weeks' gestation

OTHER OUTCOMES:
Number of oocytes retrieved | 1 month
  Number of oocytes retrieved
Fertilization rate | 1 month
  Number of 2PNs/number of inseminated M2s
Blastulation rate | 1 month
  Number of blastocysts/number of 2PNs

CONTACTS AND LOCATIONS:
Overall Officials: Jason Franasiak, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- IVI RMA New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided